CLINICAL TRIAL: NCT04985760
Title: Safety, Tolerability and Immunogenicity of Recombinant HIV Envelope Protein VRC-HIVRGP096-00-VP (Trimer 4571) Vaccine, in HIV-1 Infected Adults on Suppressive ART
Brief Title: Evaluation of Trimer 4571 Therapeutic Vaccination in Adults Living With HIV on Suppressive Antiretroviral Therapy
Acronym: NETI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Madhu Chhanda Choudhary (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Madhu Chhanda Choudhary, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIDS-ES 38763; U01AI152969 (NIH)
Record Dates: First submitted 2021-07-21; First posted 2021-08-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
Keywords: HIV; Vaccine; Vaccination; Immune system; Antibody; Antibodies; broadly neutralizing; bnabs
MeSH Terms: conditions — HIV Infections | interventions — Aluminum Hydroxide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, dose escalation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Randomized Blinded Trimer 4571 Vaccine 100mcg (Experimental): Six (6) participants will receive Trimer 4571 vaccine 100mcg with 500mcg alum adjuvant as a 1ml intramuscular injection at Day 0, Week 8 and Week 20.
  Interventions: Biological: Trimer 4571 vaccine 100mcg with 500mcg alum adjuvant
- Randomized Blinded Placebo for Trimer 4571 Vaccine 100mcg (Placebo Comparator): Two (2) participants will receive the placebo control for Trimer 4571 vaccine 100mcg as a 1ml intramuscular injection at Day 0, Week 8 and Week 20.
  Interventions: Biological: Placebo control for Trimer 4571 vaccine 100mcg with 500mcg alum adjuvant
- Randomized Blinded Trimer 4571 Vaccine 500mcg (Experimental): Eighteen (18) participants will receive Trimer 4571 vaccine 500mcg with 500mcg alum adjuvant as a 1.1ml intramuscular injection at Day 0, Week 8 and Week 20.
  Interventions: Biological: Trimer 4571 vaccine 500mcg with 500mcg alum adjuvant
- Randomized Blinded Placebo for Trimer 4571 Vaccine 500mcg (Placebo Comparator): Six (6) participants will receive the placebo control for Trimer 4571 vaccine 500mcg as a 1.1ml intramuscular injection at Day 0, Week 8 and Week 20.
  Interventions: Biological: Placebo control for Trimer 4571 vaccine 500mcg with 500mcg alum adjuvant

INTERVENTIONS:
Biological: Trimer 4571 vaccine 100mcg with 500mcg alum adjuvant — Investigational vaccine composed of Trimer 4571 100mcg, alum (aluminum hydroxide suspension) adjuvant 500mcg, and phosphate buffered saline diluent
  Other Names: HIV-1 Trimer 4571 Vaccine; VRC-HIVRGP096-00-VP
  Arms: Randomized Blinded Trimer 4571 Vaccine 100mcg
Biological: Placebo control for Trimer 4571 vaccine 100mcg with 500mcg alum adjuvant — Volume matched control for Trimer 4571 vaccine 100mcg
  Other Names: Phosphate buffered saline
  Arms: Randomized Blinded Placebo for Trimer 4571 Vaccine 100mcg
Biological: Trimer 4571 vaccine 500mcg with 500mcg alum adjuvant — Investigational vaccine composed of Trimer 4571 500mcg, alum (aluminum hydroxide suspension) adjuvant 500mcg, and phosphate buffered saline diluent
  Other Names: HIV-1 Trimer 4571 Vaccine; VRC-HIVRGP096-00-VP
  Arms: Randomized Blinded Trimer 4571 Vaccine 500mcg
Biological: Placebo control for Trimer 4571 vaccine 500mcg with 500mcg alum adjuvant — Volume matched control for Trimer 4571 vaccine 500mcg
  Other Names: Phosphate buffered saline
  Arms: Randomized Blinded Placebo for Trimer 4571 Vaccine 500mcg

SUMMARY:
Trimer 4571 is a vaccine designed to stimulate the development of broadly neutralizing antibodies (bnAbs) against HIV. Trimer 4571 is investigational, meaning it is not approved by the US Food and Drug Administration (FDA). There is limited human experience with the Trimer 4571 vaccine administered with aluminum hydroxide (alum) and the vaccine has not been tested in people with HIV prior to this study although it has been tested in healthy volunteers. The goal of this study is to see if Trimer 4571 is safe and well tolerated and to see if it will help the immune system produce bnAbs against HIV.

DETAILED DESCRIPTION:
The immune system is composed of special cells, proteins, tissues, and organs that protect against germs and microorganisms and is the body's defense against infections. Antibodies are a type of protein that helps the body fight infection and are usually made by a person's own immune system. A type of antibody that can recognize and block many types of HIV from entering healthy cells are called broadly neutralizing antibodies, or 'bnAbs', and may also activate other immune cells to help destroy HIV-infected cells. Research has shown that people with HIV who develop bnAbs against the virus are better able to control the infection. While the immune systems of some people with HIV show signs of early bnAb production, only a small percentage of people with HIV naturally develop bnAbs.

Approximately 32 participants will be sequentially enrolled and randomized 3:1 by chance like rolling dice to receive either the Trimer 4571 vaccine or a placebo vaccine that does not contain Trimer 4571.

Participants will be asked to attend 11 study visits over a period of approximately 50 weeks and receive 3 doses of their assigned study vaccine: one at Entry, one at Week 8 and one at Week 20. Researchers will compare the results from participants who get the Trimer 4571 vaccine with results from participants who get the placebo vaccine. Participants, the researchers and the clinic staff will not know which vaccine participants are getting.

After Week 20, participants will be followed for 24 additional weeks with study visits and tests to monitor their health and safety and to see how the study vaccine affects the immune system and the virus.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, documented by any FDA-approved assay. NOTE: The term 'licensed' refers to a US FDA approved kit, which is required for all investigational new drug (IND) studies.
2. Receiving continuous antiretroviral therapy (ART) for at least 24 months (defined as no interruptions longer than 30 consecutive days) and with no changes in the components of the ART for at least 8 weeks prior to study entry. A change in formulation (for example tenofovir disaproxil fumarate to tenofovir alafenamide) will not be considered a change in ART.
3. Screening CD4+ cell count ≥200cells/mm3 obtained within 60 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent.
4. Plasma HIV-1 RNA levels < 50 copies/ml for at least 24 months on ART prior to study entry using a FDA-approved assay performed by any laboratory that has a CLIA certification or its equivalent. Participants must have at least one documented HIV-1 RNA < 50 copies/ml within 12 months prior to study entry. All available HIV-1 RNA measurements must be < 50 copies/ml during the 24 months prior to study entry except as allowed by the following note.

   NOTE: Unconfirmed plasma HIV-1 RNA > 50 copies/ml but <200 copies/mL is allowed if followed by a subsequent value < 50 copies/ml.
5. Screening HIV-1 RNA levels <50 copies/mL using a FDA-approved assay performed by any laboratory that has a CLIA certification or its equivalent within 60 days prior to entry.
6. Men and women ages > 18 years.
7. The following laboratory values obtained within 60 days prior to entry:

   * Hemoglobin ≥10 g/dL
   * Absolute neutrophil count (ANC) ≥1000/mm3
   * Platelet count ≥100,000/mm3
   * Creatinine ≤ 1.5x upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) (SGPT) ≤2.5x ULN
8. Ability and willingness of participant to provide informed consent.
9. In the opinion of the investigator, no medical, mental health or other condition that precludes participation.
10. For persons who can become pregnant, negative serum or urine pregnancy test within 48 hours prior to entry by any US clinic or laboratory that has a CLIA certification or its equivalent, or is using a point-of-care (POC)/ CLIA-waived test. Persons who can become pregnant include women who have not been post-menopausal for at least 12 consecutive months, (i.e., who have had menses within the preceding 12 months) or women who have not undergone surgical sterilization (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation or salpingectomy). Self- report is acceptable documentation of menopause and sterilization.
11. All participants must agree not to participate in the conception process (eg, active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the participant/partner must use at least one reliable form of contraception (condoms, with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an IUD; or hormone-based contraceptive), while receiving study treatment and for 12 weeks following the final study vaccine.

Exclusion Criteria:

1. Known to have been started on antiretroviral therapy within 3 months of the presumed or known date of first acquiring HIV-1 infection; i.e., treated during acute HIV-1 infection
2. Currently breastfeeding or pregnant
3. Known allergy/sensitivity or any hypersensitivity to components of study vaccine or their formulation.
4. Known chronic inflammatory conditions such as, but not limited to, rheumatoid arthritis, systemic lupus erythematosus, sarcoidosis, inflammatory bowel disease (i.e., Crohn's disease or ulcerative colitis), chronic pancreatitis, or autoimmune hepatitis, myositis, or myopathy.
5. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
6. Serious medical illness that requires systemic treatment and/or hospitalization within 30 days prior to entry.
7. Use of systemic immunomodulators (e.g., interleukins, interferons, Cyclosporine), systemic cytotoxic chemotherapy, or investigational therapy within 60 days prior to study entry.

   NOTE: Participants receiving stable physiologic doses of glucocorticoids, defined as the equivalent of prednisone ≤10 mg/day, will not be excluded. Stable physiologic glucocorticoid doses should not be discontinued for the duration of the study. In addition, participants receiving inhaled or topical corticosteroids, or topical imiquimod will not be excluded.
8. Receipt of any investigational HIV immunotherapy or HIV therapeutic vaccination within 12 months prior to study entry.
9. History of positive HCV antibody with detectable HCV RNA in plasma within 48 Weeks prior to study entry. NOTE: Persons with positive HCV Ab but negative plasma HCV RNA are allowed to participate. Sites must document negative HCV RNA within 24 weeks of study entry.
10. Treatment for hepatitis C within 6 months prior to study entry.
11. History of positive HBsAg within 48 weeks prior to study entry.
12. History of severe reaction or anaphylaxis to prior vaccinations.
13. Body Mass Index >40kg/m2.
14. Receipt of Blood products or immune globulins within 16 weeks prior to Enrollment as per protocol section 5.3.2.
15. Receipt of Live attenuated vaccines within 4 weeks prior to enrollment.
16. Current allergen immunotherapy with antigen injections, unless on maintenance schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of three vaccinations of Trimer 4571 vaccine in adults with HIV on suppressive ART | Day 0 through Week 44
  The proportion of participants experiencing at least one Grade 3 or higher adverse event will be summarized within and across the Trimer 4571 vaccine 100mcg, Trimer 4571 vaccine 500mcg and placebo control vaccine groups. The number of adverse events in each group will also be summarized by severity, body system, and relationship to study vaccine using frequencies, percent, and 95% confidence intervals.

SECONDARY OUTCOMES:
Immunogenicity of three vaccinations of Trimer 4571 vaccine in adults with HIV on suppressive ART | Baseline and Week 22
  Comparison of the change in the serum ID50 neutralization titer of BG505.W6M.C2 virus between Trimer 4571 vaccine 100mcg, Trimer 4571 vaccine 500mcg, and placebo control vaccine. Vaccine responders will be as defined by either (i) 4-fold increase in neutralization titer from pre-vaccination to at least one virus in the curated virus panel at any protocol-specified time point post vaccination and/or (ii) Evidence of BG505.W2 neutralization at any protocol-specified time point post vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Madhu Choudhary, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - AIDS Clinical Trials Unit/The Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No